CLINICAL TRIAL: NCT05656274
Title: A Phase 1b，Randomized, Investigator/Participant-Blind, Placebo-Controlled, Multiple-Ascending Dose Trial to Evaluate the Safety, Tolerance and Pharmacokinetics of JS1-1-01 in Healthy Subjects
Brief Title: A Study of the Safety,Tolerability,and Pharmacokinetics of Multiple-Ascending Dose JS1-1-01 in Healty Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: TSL-CM-JS1-1-01-Ⅰb
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JS1-1-01 (Experimental): JS1-1-01 25mg，50mg，100mg，150mg
  Interventions: Drug: JS1-1-01
- Placebo (Placebo Comparator): placebo 25mg，50mg，100mg，150mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JS1-1-01 — Oral tables
  Arms: JS1-1-01
Drug: Placebo — Oral tables
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety，tolerability，and pharmacokinetics of multiple-accending dose of JS1-1-01。

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants 18 to 45 years of age.
2. Body weight ≥ 50 kg ; body mass index of 19 to 28 kg/m^2 ;
3. Subjects have no birth plan and voluntarily take effective contraceptive measures within 3 months after signing the informed consent form and the last medication;
4. Willing and able to sign the informed consent form, and understand and abide by the research procedures.

Exclusion Criteria:

1. Allergic constitution or a history of food and drug allergy;
2. According to the Columbia Suicide Severity Scale (C-SSRS), subjects have suicide risk , or have a history of self mutilation;
3. There are neurological/psychiatric, respiratory, cardiovascular, gastrointestinal, blood and lymphatic, endocrine, skeletal and muscular diseases, liver and kidney dysfunction, or any other diseases and physiological conditions that may affect the study;
4. The results of vital signs, physical examination, electrocardiogram and laboratory examination are abnormal and clinically significant;
5. HBsAg, HCV antibody, HIV antibody or Treponema pallidum specific antibody were positive;
6. Pregnant or lactating women;
7. A History of drug abuse, or positive urine drug abuse screening;
8. Smoking more than 5 cigarettes per day in the last 3 months, or not completely quitting smoking during the study period;
9. In recent three months, the amount of alcohol consumed per week exceeded 14 units of alcohol , or the alcohol breath test was positive, or alcohol consumption was prohibited from 48 hours before the first administration to the end of the test;
10. Those who have taken any drugs within 4 weeks before the first administration (including prescription drugs, over-the-counter drugs, Chinese herbal medicine, vitamins, calcium tablets and other food supplements);
11. Difficulty in blood collection and history of blood sickness and needle sickness;
12. Those who have special requirements on diet and can not follow the unified diet, or are prone to diarrhea, nausea, vomiting, abdominal distension or other gastrointestinal discomfort after drinking milk or dairy products;
13. From 48 hours before the first administration to the end of the study, the subjects refused to stop using any drink or food containing methylxanthine, such as coffee, tea, cola, chocolate, etc;
14. From 7 days before the first administration to the end of the study, the subjects refused to stop using any drink or food containing grapefruit;
15. Participated in any drug clinical trial and took the test drug in recent 3 months; Or those who plan to participate in other clinical trials during the trial
16. Those who have donated blood or lost blood ≥ 200 mL or received blood transfusion or used blood products in recent 3 months; Or those who plan to donate blood during the trial;
17. The researchers believe that the subjects have poor compliance or other clinical, social or family factors that are not suitable for inclusion.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | day 11
  To evaluate the safety and tolerability of JS1-1-01 in healthy participants by assessing the number, severity and type of adverse events, including changes in laboratory safety tests and electrocardiogram (ECG)

SECONDARY OUTCOMES:
Pharmacokinetics profile after a single dose | day 1
  Cmax of JS1-1-01 and its major metabolites after a single dose.
Pharmacokinetics profile after a single dose | day 1
  Tmax of JS1-1-01 and its major metabolites after a single dose.
Pharmacokinetics profile after a single dose | day 1
  t1/2 of JS1-1-01 and its major metabolites after a single dose.
Pharmacokinetics profile after a single dose | day 1
  AUC0-t of JS1-1-01 and its major metabolites after a single dose.
Pharmacokinetics profile after a single dose | day 1
  AUC0-∞ of JS1-1-01 and its major metabolites after a single dose.
Pharmacokinetics profile after a single dose | day 1
  λz of JS1-1-01 and its major metabolites after a single dose.
Pharmacokinetics profile after a single dose | day 1
  Vd/F of JS1-1-01 and its major metabolites after a single dose.
Pharmacokinetics profile after a single dose | day 1
  CL/F of JS1-1-01 and its major metabolites after a single dose.
Pharmacokinetics profile after multiple dosing. | day 11
  Css_min of JS1-1-01 and its major metabolites after multiple dosing.
Pharmacokinetics profile after multiple dosing. | day 11
  Css_max of JS1-1-01 and its major metabolites after multiple dosing.
Pharmacokinetics profile after multiple dosing. | day 11
  Css_av of JS1-1-01 and its major metabolites after multiple dosing.
Pharmacokinetics profile after multiple dosing. | day 11
  AUC0-tau of JS1-1-01 and its major metabolites after multiple dosing.
Pharmacokinetics profile after multiple dosing. | day 11
  AUC0-∞,ss of JS1-1-01 and its major metabolites after multiple dosing.
Pharmacokinetics profile after multiple dosing. | day 11
  AUC0-t,ss of JS1-1-01 and its major metabolites after multiple dosing.
Pharmacokinetics profile after multiple dosing. | day 11
  Tmax,ss of JS1-1-01 and its major metabolites after multiple dosing.
Pharmacokinetics profile after multiple dosing. | day 11
  T1/2,ss of JS1-1-01 and its major metabolites after multiple dosing.
Pharmacokinetics profile after multiple dosing. | day 11
  CLss/F of JS1-1-01 and its major metabolites after multiple dosing.
Pharmacokinetics profile after multiple dosing. | day 11
  DF of JS1-1-01 and its major metabolites after multiple dosing.
Pharmacokinetics profile after multiple dosing. | day 11
  Rac of JS1-1-01 and its major metabolites after multiple dosing.

OTHER OUTCOMES:
Pharmacodynamics：Concentration of BDNF | day 9
  Concentration of BDNF(Brain derived neurotrophic factor)
Pharmacodynamics：Changes in heart rate and blood pressure | day 9
  Changes in heart rate and blood pressure (systolic/diastolic) compared with baseline
Pharmacodynamics：Incidence of AESI | day 11
  Incidence of AESI（adverse event of special interest） (nausea, dry mouth, headache, sweating, somnolence)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, China